CLINICAL TRIAL: NCT06144398
Title: Single Use Versus Standard Flexible Bronchoscopes in Interventional Pulmonary Procedures: an Open Label Randomized Controlled Trial
Brief Title: Single Use Flexible Bronchoscopes in Interventional Pulmonary Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Goran Glodić, MD, Principal Investigator, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8.1-22/21-2; 02/013AG
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Atelectasis; Hemoptysis; Stridor
Keywords: Bronchoscopy; Single Use Flexible Bronchoscope; Interventional Pulmonology
MeSH Terms: conditions — Pulmonary Atelectasis; Hemoptysis; Respiratory Sounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Use Bronchoscope (Experimental)
  Interventions: Device: Single Use Bronchoscope
- Standard Bronchoscope (Active Comparator)
  Interventions: Device: Standard Bronchoscope

INTERVENTIONS:
Device: Single Use Bronchoscope — The interventional procedure is performed with a single use bronchoscope.
  Arms: Single Use Bronchoscope
Device: Standard Bronchoscope — The interventional procedure is performed with a standard bronchoscope.
  Arms: Standard Bronchoscope

SUMMARY:
Single Use Flexible bronchoscopes have gained popularity in recent years and are becoming technologically more advanced. They are widely accepted and used in everyday practice for simple procedures. The aim of this study is to evaluate single use flexible bronchoscopes in more advanced settings, such as interventional pulmonary procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients requiring an interventional pulmonary procedure during the study period
* Signed informed consent

Exclusion Criteria:

* Any patient with a contraindication for rigid and/or flexible bronchoscopy
* Coagulopathy (PV INR > 1.3)
* Thrombocytopenia (<50x10*9 or anemia (Hgb <80 g/L)
* DOAC, LMWH or antiplatelet drug therapy
* Thrombophilia, history of pulmonary embolism or deep vein thrombosis
* Contraindication for endobronchial application of adrenaline
* Uncontrolled coronary artery disease, cerebrovascular disease or arrhythmia
* Uncontrolled pulmonary hypertension
* Cardiovascular decompensation
* Severe hypoxia (PaO2 <60mmHg, SaO2 <90% with an FiO2 >=60%)
* Cervical spine instability

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Overall performance | through study completion, an average of 12 months
  Overall performance of the bronchoscope as graded by the operator (on a scale from 1 to 10; 1 worse, 10 best performance)

SECONDARY OUTCOMES:
Functionality, handle and interface | through study completion, an average of 12 months
  Functionality, handle and interface of the bronchoscope as graded by the operator (on a scale from 1 to 10; 1 worse, 10 best performance)
Suction | through study completion, an average of 12 months
  Suction power of the bronchoscope as graded by the operator (on a scale from 1 to 10; 1 worse, 10 best performance)
Image quality | through study completion, an average of 12 months
  Image quality as graded by the operator (on a scale from 1 to 10; 1 worse, 10 best performance)
Bleeding control | through study completion, an average of 12 months
  Bleeding control as graded by the operator (on a scale from 1 to 10; 1 worse, 10 best performance)
Compatibility | through study completion, an average of 12 months
  Compatibility with other devices (i.e. ballon blockers, forceps, laser, cryprobe) as graded by the operator (on a scale from 1 to 10; 1 worse, 10 best performance)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia